CLINICAL TRIAL: NCT01656421
Title: Assessment of Risk in Chronic Airways Disease Evaluation (ARCADE)
Brief Title: Assessment of Risk in Chronic Airways Disease Evaluation
Acronym: ARCADE
Status: Completed | Type: Observational
Sponsor: Cardiff University (Other)
Collaborators: GlaxoSmithKline (Industry); Cardiff Metropolitan University (Other)
Responsible Party: Principal Investigator, Nichola Gale, Lecturer, Cardiff University
Other Study IDs: SPON 87610; 10/CAD/4972 (Other: Cardiff & Vale UHB R&D Office)
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD: Patients with Chronic Obstructive Pulmonary Disease, including mild, moderate, severe and very severe airflow obstruction
- Comparators: Current or ex-smokers free from from Respiratory Disease

SUMMARY:
Patients with chronic obstructive pulmonary disease (COPD) have an increased risk of cardiovascular disease,osteoporosis, muscle wasting and diabetes mellitus. Cardiovascular disease is a major cause of death in such patients and it may be related to excess stiffening of the walls of major arteries, such as the aorta, and it has been suggested to represent premature aging. However, there is little known of the development of these problems, which were previously considered to be due to smoking and which is now known not to be the only factor. The investigators will study a large group of patients with mild to very severe airflow obstruction based on the NICE 2010 classification of severity and a matched comparator group free of COPD. This study involves three assessments of the development of the complications of COPD over a five year period. The key measure will be the rate of change in the aortic wall stiffness, an accepted indicator of the risk of heart disease. Changes in wall stiffness will be related to the severity of lung disease; other known cardiovascular risk factors, such as high blood pressure, increased blood cholesterol and to cardiovascular events including heart attacks and death; and to the presence of other complications, such as osteoporosis, muscle wasting and diabetes mellitus. These measures will be analysed in the context of changes in bodywide inflammation and metabolic function and the changes in the rate of ageing. This increased knowledge of interacting factors in the complications of COPD is likely to lead to studies of treatments to avoid their development.

ELIGIBILITY:
Inclusion Criteria:

* Previously Proven COPD or at risk of developing COPD

Exclusion Criteria:

* Pregnancy
* A history of malignancy in the last 5 years
* Unable to give informed consent or diagnosed dementia
* Renal or hepatic failure
* Active endocrine disorder eg., Addison's disease, hypothyroidism
* Any other disease identified as having an inflammatory or metabolic component, eg. rheumatoid disease
* Disorders affecting mobility, eg. Parkinson's disease, cerebrovascular accident.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 767 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Aortic Pulse Wave Velocity (arterial stiffness) | Baseline, 2 and 5 yrs
  Rate of change in aortic pulse wave velocity in patients with COPD over a period of 5 years and its relationship to cardiovascular morbidity and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Barry J McDonnell, PhD BSc, Principal Investigator — Cardiff Metropolitan University; John R Cockcroft, MD, FRCP, Study Chair — Cardiff Metropolitan University
Locations (1):
- Cardiff Metropolitan University, Cardiff, United Kingdom

REFERENCES:
- [Derived] Mohan D, Forman JR, Allinder M, McEniery CM, Bolton CE, Cockcroft JR, MacNee W, Fuld J, Marchong M, Gale NS, Fisk M, Nagarajan S, Cheriyan J, Lomas DA, Calverley PMA, Miller BE, Tal-Singer R, Wilkinson IB, Polkey MI; ERICA Consortium. Fibrinogen does not relate to cardiovascular or muscle manifestations in COPD: cross-sectional data from the ERICA study. Thorax. 2018 Dec;73(12):1182-1185. doi: 10.1136/thoraxjnl-2018-211556. Epub 2018 Apr 4. PMID 29618495
- [Derived] Gale NS, Albarrati AM, Munnery MM, Munnery IC, Irfan M, Bolton CE, Rambaran CN, Singer RM, Cockcroft JR, Shale DJ. Assessment of Risk in Chronic Airways Disease Evaluation (ARCADE): Protocol and preliminary data. Chron Respir Dis. 2014 Nov;11(4):199-207. doi: 10.1177/1479972314546765. Epub 2014 Aug 26. PMID 25159833